CLINICAL TRIAL: NCT04954066
Title: Association Between Muscular Tissue Oxygen Saturation and Postoperative Acute Kidney Injury in Older Patients Undergoing Major Abdominal Surgery: A Prospective Cohort Study
Brief Title: Association Between Muscular Tissue Oxygen Saturation and AKI in Older Patients Undergoing Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: lingzi-2021-1; Yinlingzi (Registry Identifier: Yinlingzi)
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-08

CONDITIONS: Acute Kidney Injury
Keywords: postoperative acute kidney injury; muscular tissue oxygen saturation; Near-infrared spectroscopy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate association between muscular oxygen saturation and postoperative acute kidney injury(AKI) in older patients undergoing abdominal surgeries.The investigator also intend to explore the thresholds of muscular oxygen saturation that correlate with a reduced risk of AKI and therefore have the potential to be used as therapeutic targets in future.

DETAILED DESCRIPTION:
Acute kidney injury is one of the common and serious complications after major abdominal surgeries,which a reported incidence is as high as 7.5-13.4%.The evidence shows that nearly 20% of elder patients with comorbidity are severely related to postoperative AKI,which lead to increased complications, prolonged stays in hospital and higher mortality.What'more,even smaller increases in the levels of serum creatinine (sCr) may predict worse kidney function after 1or 2 years.But there is no effective treatment or strategy for acute kidney injury at the moment.Therefore,early identification and prevention for AKI in perioperative period are key points.

The mechanism of AKI is complex and multifaceted,which includes that surgeries or anesthesia lead to renal hypoperfusion,ischemia and hypoxia. If the anesthesiologists can monitor the oxygenation status of renal tissues and improve it during surgery, it may reduce the incidence of AKI.

Near-infrared spectroscopy (NIRS) is a new noninvasive technique that continuously monitors tissue oxygen saturation by measuring the relative concentrations of oxygenated and deoxygenated hemoglobin within a local tissue area.It has been improved that perioperative muscular oxygen saturation is related to patients outcome.A observational study showed an association between lower intraoperative tissue oxygen saturation monitored on both sides of paraspinal muscle and higher risk of postoperative AKI in patients having cardiac surgery, suggesting a potential similarity of tissue perfusion and oxygenation between renal and muscular tissue beds.

Therefore,in this study, the investigator hypothesizes that monitoring muscular oxygen saturation during period may reflect some part of renal tissue oxygen saturation and associate with postoperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old,
* ASA scoreⅠ-Ⅲ,
* Scheduled to undergo a 2-hour-or-longer elective major abdominal surgeries

Exclusion Criteria:

* Urological surgery or procedure related to renal tissue may be performed during surgeries.
* Nephrectomy or partial nephrectomy was performed before surgeries.
* Preoperative glomerular filtration rate<30ml/1.73m2, or end-stage renal disease or renal transplant.
* Poor hearing or vision and language barrier impeding postoperative assessment.
* Skin condition incompatible with the adhesive oximetry probe.
* Refuse to participate in the trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study intend to enroll elder patients having major abdominal surgeries in our center.
Sampling Method: Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
the incidence of AKI in 7 days | All the patients will be observed in previous 7 days after surgery for AKI.
  Postoperative AKI will be diagnosed according to KDIGO(Kidney Disease Improving Global)as one of the following:
  An increase in serum creatinine by≥0.3 mg/dl ( ≥26.5μmol/l) within 48 h; An increase in serum creatinine to ≥1.5 times baseline within the previous 7 days; Urine volume≤0.5 ml/kg/h for 6 h.

SECONDARY OUTCOMES:
the incidence of other complications,hospital stays and mortality in 30 days | All the patients will be followed up within 30 days after surgery.
  It includes cardio-cerebrovascular complications,pneumonia,infection,unplanned transfer to ICU,ICU stays and other dysfunction.The severity of complications was categorised as mild,moderate, severe, or fatal using a modified Clavien-Dindo classification.
  scheme.

CONTACTS AND LOCATIONS:
Overall Officials: N xinli, MD, Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No